CLINICAL TRIAL: NCT02196571
Title: The Impact of Structured Aerobic and Resistance Exercise on the Course and Outcome of Gestational Diabetes Mellitus
Brief Title: Structured Aerobic and Resistance Exercise and Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association for Functional Rehabilitation, Recreation and Applied Kinesiology Impulse (Other)
Responsible Party: Principal Investigator, Iva Sklempe Kokic, PT, PgD Kin, Association for Functional Rehabilitation, Recreation and Applied Kinesiology Impulse
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Impuls001
Record Dates: First submitted 2014-07-19; First posted 2014-07-22 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Gestational Diabetes Mellitus
Keywords: GDM; Exercise; Diabetes; Pregnancy
MeSH Terms: conditions — Diabetes, Gestational; Motor Activity; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise and lifestyle change (Experimental): Women in the experimental group will be included in structured exercise programme two times per week with duration of 50 minutes.Participants will start with training sessions right after they are diagnosed with GDM and they will exercise until the end of the pregnancy or occurence of contraindications. Programme will consist of aerobic exercises (20 minutes), resistance exercises (20 minutes), plevic floor, stretching and relaxation exercises (10 minutes). Women in control group will receive standard antenatal care.
  Interventions: Other: Structured Exercise
- Control (No Intervention): Standard antenatal care

INTERVENTIONS:
Other: Structured Exercise
  Arms: Exercise and lifestyle change

SUMMARY:
Gestational diabetes mellitus (GDM) is defined as impaired glucose tolerance of various degrees first manifested during pregnancy. The primary aim of treating GDM is to optimize glycaemic control and improve pregnancy outcomes. Also, as part of treatment, it is recommended to continue or initiate exercising with moderate intensity. However, available data on the effects of physical activity on GDM are based on a small number of trials. The aim of the trial is to examine and add new scientific evidence on possible health-related effects of application of structured programme consisting of aerobic and resistance exercises on the course and outcomes of GDM. Primary goal of research is to determine how proposed exercise programme effects glycaemic control, rate of complications during pregnancy, labour, delivery, immediate after delivery and health status of newborn. Main hypothesis is that parameters of glycaemic control, course of GDM, complications during delivery and birth outcomes directly and significantly correlate with participation in structured programme of exercise. Research will be conducted as experimentally designed randomized controlled trial. Participants will be pregnant women diagnosed with GDM, age between 20 and 40, without comorbidities. Women in the experimental group will be included in exercise programme two times per week with duration of 50 minutes. Training sessions will start right after the diagnosis and will be performed until the end of the pregnancy. The training protocol will follow international guidelines (ACOG, 2001; ACOG, 2002; ADA, 2008; NICE, 2008; ADA 2011). Women in the control group will receive standard medical care.

ELIGIBILITY:
Inclusion Criteria:

* established diagnosis of gestational diabetes,
* age between 20 and 40,
* otherwise healthy pregnancy

Exclusion Criteria:

* pharmacological treatment with oral hypoglicemics and/or insulin therapy introduced prior to trial enrollment,
* existing comorbidities and
* contraindications for exercise

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of pregnant women with complications during pregnancy, labour and delivery | up to labour
  Blood glucose levels, need for insulin and oral hypoglycemic drugs, need for cesarean section and other operative delivery methods, other adverse occurences during pregnancy, labour and delivery

SECONDARY OUTCOMES:
Number of macrosomic infants | delivery
Weight gain in pregnancy | After recruitment and during pregnancy (30, 33 and 36 weeks)
  Body mass and percentage of fat measured by caliper

OTHER OUTCOMES:
Low Back Pain | after recruitment and during pregnancy (30 and 36 weeks)
  Visual analogue scale Roland-Morris Low Back Pain and Disability Questionnaire Pelvic Girdle Questionnaire
Physical Activity in Pregnancy | After recruitment and in 30th and 36th week of pregnancy
  Pregnancy Physical Activity Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Iva Sklempe Kokic, PT, PgD Kin, Principal Investigator — Association for functional rehabilitation, recreation and applied kinesiology Impuls
Locations (1):
- Association for functional rehabilitation, recreation and applied kinesiology Impuls, Zagreb, Croatia